CLINICAL TRIAL: NCT02808117
Title: Microfinance Institutions as a Platform for Global Health Delivery: Evidence From a Pilot Program
Brief Title: Microfinance Institutions as a Platform for Global Health
Status: Completed | Type: Observational
Sponsor: Columbia University (Other)
Responsible Party: Principal Investigator, Aaron Isaac Baum, Co-Investigator, Columbia University
Other Study IDs: AAAP7004
Record Dates: First submitted 2016-06-17; First posted 2016-06-21 (Estimated); Last update posted 2016-11-30 (Estimated); Status verified 2016-11

CONDITIONS: Malnutrition; Anemia
Keywords: microfinance institution; MFI
MeSH Terms: conditions — Malnutrition; Anemia

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Targeted initially: Children who were in the Haiti villages and targeted by the MFI program with MNP delivery initially.
  Interventions: Dietary Supplement: MNP
- Targeted later: Children who were in the Haiti villages and not targeted by the MFI program with MNP delivery until later.
  Interventions: Dietary Supplement: MNP

INTERVENTIONS:
Dietary Supplement: MNP — Program that delivered MNP and implemented by an MFI in Haiti during 2011-2012.
  One form of micronutrient supplementation proven to effectively combat micronutrient deficiency.
  Other Names: Micronutrient powders; Sprinkles

SUMMARY:
This study will analyze data from a program run by an microfinance institution (MFI) in Haiti from 2011-2012 where the MFI delivered health goods to some of the villages where it operates. By comparing health indicators among children who were in villages targeted by the program initially to children who were in villages that were not targeted by the program until later, the investigators hope to understand if the MFI successfully delivered the intervention and offer a practical platform for delivery of basic health goods.

DETAILED DESCRIPTION:
Two-thirds of child deaths could be prevented with increased coverage of existing health products and services; however, effectively delivering health products and services to rural populations in low-income countries remains a practical challenge. This study investigates whether microfinance institutions (MFIs), having invested in community-based infrastructure to deliver financial services to 200 million rural poor households globally, offer a practical platform for delivery of basic health goods.

The investigators intend to analyze data from a pilot program implemented by an MFI in Haiti during 2011-2012 that distributed an evidence-based health good, micronutrient powders (MNPs), to 526 children in 34 villages where the MFI operates. Micronutrient deficiency is estimated to be responsible for over 1 million deaths of children under five per year. MNPs are one form of micronutrient supplementation proven to effectively combat micronutrient deficiency.

Published cost estimates indicate that leveraging existing supply chains could cut the total cost of mass MNP delivery by 25%. Given MFIs reach 200 million households globally, MFI-based delivery of health goods may be a promising route to improving health outcomes efficiently.

ELIGIBILITY:
Inclusion Criteria:

* Lives in a household where the head of household was an microfinance client.

Exclusion Criteria:

* Severely anemic (Hgb < 70 g/L)
* Severely malnourished (Mid Upper Arm Circumference < 110 mm)

Ages: 6 Months to 54 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Children aged 6-54 months who lived in a household where the head of household was an microfinance client.
Sampling Method: Non-Probability Sample
Enrollment: 526 (Actual)
Dates: Start 2015-05; Primary Completion 2016-08 (Actual); Study Completion 2016-11 (Actual)

PRIMARY OUTCOMES:
Change in blood hemoglobin concentration | Baseline, 3 months

SECONDARY OUTCOMES:
Prevalence of diagnosis of anemia | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Aaron I Baum, PhD, Study Director — Columbia University
Locations (1):
- Columbia University, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Undecided